CLINICAL TRIAL: NCT00000257
Title: Effects of Alcohol History on Effects of Nitrous Oxide
Brief Title: Effects of Alcohol History on Effects of Nitrous Oxide - 9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double
Other Study IDs: NIDA-08391-9; R01DA008391 (NIH); R01-08391-9
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Alcohol-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; subjective effects; ethanol; healthy volunteer
MeSH Terms: conditions — Alcohol-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Light drinkers (Active Comparator)
  Interventions: Drug: 0% N2O and 10% N2O; Drug: 0% N2O and 20% N2O; Drug: 0% N2O and 30% N2O; Drug: 0% N2O and 40% N2O
- Moderate drinkers (Active Comparator)
  Interventions: Drug: 0% N2O and 10% N2O; Drug: 0% N2O and 20% N2O; Drug: 0% N2O and 30% N2O; Drug: 0% N2O and 40% N2O

INTERVENTIONS:
Drug: 0% N2O and 10% N2O
Drug: 0% N2O and 20% N2O
Drug: 0% N2O and 30% N2O
Drug: 0% N2O and 40% N2O

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. Comparisons between nitrous oxide, opiates, and benzodiazepine antagonists will be made. To determine effects of alcohol history on the reinforcing, subjective and psychomotor effects of nitrous oxide in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 1995-09; Primary Completion 1997-04 (Actual); Study Completion 1997-04 (Actual)

PRIMARY OUTCOMES:
Choice of nitrous oxide vs placebo | After 30 min inhalation each of N2O and placebo
  Two subject groups (light drinkers vs moderate drinkers) were asked to inhale a given conc of N2O and inhale a placebo, then choose for a third inhalation. The subject & the technician administering the inhalant were blinded. Testing was done at each dose.

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Cho AM, Coalson DW, Klock PA, Klafta JM, Marks S, Toledano AY, Apfelbaum JL, Zacny JP. The effects of alcohol history on the reinforcing, subjective and psychomotor effects of nitrous oxide in healthy volunteers. Drug Alcohol Depend. 1997 Apr 14;45(1-2):63-70. doi: 10.1016/s0376-8716(97)01346-x. PMID 9179508